CLINICAL TRIAL: NCT04629911
Title: The Effect of High Flow Nasal Oxygenation on Gastric Insufflation in Paralyzed Anesthetized Patients Undergoing Laryngologic Surgery
Brief Title: High Flow Nasal Oxygenation and Gastric Insufflation in Anesthetized Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jong Yeop Kim, Professor, Ajou University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MED-DE1-20-424
Record Dates: First submitted 2020-11-10; First posted 2020-11-16 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Gastric Distention
MeSH Terms: interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HFNO arm (Experimental): Patients will receive HFNO therapy during laryngomicrosurgery.
  Interventions: Device: THRIVE

INTERVENTIONS:
Device: THRIVE — Patients will receive HFNO therapy during laryngomicrosurgery. Patients will undergo a gastric ultrasound examination after HFNO therapy.
  Other Names: Optiflow

SUMMARY:
Transnasal humidified rapid-insufflation ventilatory exchange(THRIVE), or also termed high flow nasal oxygenation (HFNO) is a method of supplying heated, humidified high concentrations of oxygen via nasal cavity.

The purpose of this study is to investigate the effect of HFNO on gastric insufflation in paralyzed anesthetized patients undergoing laryngologic surgery.

DETAILED DESCRIPTION:
HFNO can be used during intraoperative period. HFNO reduces the risk of desaturation and prolongs the safe apnea time, compared with conventional oxygenation.

In laryngeal microsurgery, HFNO therapy make possible to perform tubeless anesthesia, providing perfect exposure of structure of the vocal cords.

HFNO have a risk for low level of positive pressure can make gastric distension, but gastric reflux or aspiration were not occurred during rapid sequence induction for emergency operation.

The purpose of this study is to investigate the effect of HFNO on gastric insufflation in paralyzed anesthetized patients undergoing laryngologic surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology physical status classification I and II
* Patients scheduled for laryngeal microsurgery under general anesthesia

Exclusion Criteria:

* gastroesophageal reflux
* gastric pathology
* pregnancy
* major cardiovascular, pulmonary, or cerebrovascular disease
* severe obesity (body mass index>35 kg/m2)

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
change of gastric volume | before HFNO application (baseline), immediately after HFNO application
  Ultrasound exam will measure the antral cross-sectional area of gastric antrum

CONTACTS AND LOCATIONS:
Locations (1):
- Ajou University Hospital, Suwon, Gyeongki-do, South Korea